CLINICAL TRIAL: NCT01448031
Title: A Phase I, Open-label, Randomized, Two Way Crossover Pharmacokinetic Study Comparing the Bioavailability of Acetylsalicylic Acid (ASA) After 5 Days Repeated Once Daily Administration of a Fixed Dose Combination Capsule of ASA 81 mg/Esomeprazole 20 mg and ASA 80 mg (European Aspirin Reference Product)
Brief Title: A Healthy Female and Male Volunteers Aspirin Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: D961FC00012
Record Dates: First submitted 2011-09-22; First posted 2011-10-07 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Acetyl Salicylic Acid; Bioavailability; Healthy Volunteers
MeSH Terms: interventions — Esomeprazole

ARMS (2):
- 1 (Experimental): Capsule ASA 81mg/esomeprazole 20mg
  Interventions: Drug: Capsule ASA 81mg/esomeprazole 20mg
- 2 (Active Comparator): ASA (Acetylsalicylzuur Apotex cardio 80 mg) Tablet 80 mg
  Interventions: Drug: Acetylsalicylzuur Apotex Cardio

INTERVENTIONS:
Drug: Capsule ASA 81mg/esomeprazole 20mg — Multiple doses administered on Day 1 to 5
  Arms: 1
Drug: Acetylsalicylzuur Apotex Cardio — Multiple doses administered on Day 1 to 5
  Arms: 2

SUMMARY:
This is a study to compare the bioavailability of Acetyl Salicylic Acid (ASA) between Esomeprazole and Aspirin after multiple dose administration.

DETAILED DESCRIPTION:
A Phase I, open-label, randomized, two way crossover pharmacokinetic study comparing the bioavailability of acetylsalicylic acid (ASA) after 5 days repeated once daily administration of a fixed dose combination capsule of ASA 81 mg/esomeprazole 20 mg and ASA 80 mg (European aspirin reference product).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 20 to 50 years inclusive.
* Have a body body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive and weigh 50.0 to 100.0 kg inclusive.
* Females must be of non-childbearing potential or be of childbearing potential but have a negative serum hCG pregnancy test during screening and on admission.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study.
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the Investigator.
* History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic profile of acetylsalicylic acid (ASA) and salicylic acid (SA) in terms of area under curve (AUC), maximum concentration at steady state (Css,max), time to reach maximum concentration (tmax) and terminal half- time (t1/2). | Day 5
  PK samples collected pre-dose and at 5mins, 10 mins, 20 mins, 30 mins, 40mins, 50 mins, 1hr 15 mins, 1.5hrs, 2 hrs, 2hr 30 mins, 3hrs, 3hr 30 mins, 4 hrs, 5 hrs, 6hrs, 8hrs,10 hrs, 12hrs post-dose.

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events, blood pressure, pulse, ECG (Electrocardiogram), physical examination, safety labs | Pre-dose up to 7 day after last dose
  No formal statistical tests will be performed. Abnormalities will be listed without statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Beboso, Principal Investigator — BioKinetic Europe Ltd,14 Great Victoria Street,Belfast, N.Ireland,United Kingdom BT2 7BA; Tore Lind, Study Director — AstraZeneca, Pepparedsleden 1 431 83 Molndal Sweden
Locations (1):
- Research Site, London, UK, United Kingdom